CLINICAL TRIAL: NCT05484908
Title: Efficacy and Safety of Artificial Liver Support System Treatment for Immune Checkpoint Inhibitors Related Liver Failure in Patients With Hepatocellular Carcinoma
Brief Title: Efficacy and Safety of ALSS Treatment for ICIs-LF in Patients With HCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Wenxiong Xu, Associate Chief Physician, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XWX4
Record Dates: First submitted 2022-07-30; First posted 2022-08-02 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Immune-Mediated Hepatitis; Liver Failure; Hepatocellular Carcinoma
MeSH Terms: conditions — Liver Failure; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DPMAS+LPE group (Experimental): 30 patients receive treatment of DPMAS, LPE, and comprehensive internal medical treatment.
  Interventions: Other: DPMAS+LPE; Other: Comprehensive internal medical treatment
- PE group (Active Comparator): 30 patients receive treatment of PE and comprehensive internal medical treatment.
  Interventions: Other: PE; Other: Comprehensive internal medical treatment

INTERVENTIONS:
Other: DPMAS+LPE — Patients will receive treatment of double plasma molecular adsorption system (DPMAS) and low volume plasma exchange (LPE) for three times in two weeks. The volume of plasma adsorption in DPMAS is 5000~6000 millilitre. The volume of fresh frozen plasma used in LPE is 1000 millilitre.
  Arms: DPMAS+LPE group
Other: PE — Patients will receive treatment of plasma exchange (PE) for three times in two weeks. The volume of fresh frozen plasma used in PE is 2000 millilitre.
  Arms: PE group
Other: Comprehensive internal medical treatment — Patients will receive comprehensive internal medical treatment.

SUMMARY:
This study aims to investigate the efficacy and safety of artificial liver support system treatment for immune checkpoint inhibitors related liver failure in patients with hepatocellular carcinoma.

DETAILED DESCRIPTION:
Immune checkpoint inhibitors (ICIs) are commonly used for advanced stage of hepatocellular carcinoma (HCC) in recent years. The incident rate of Grade 4 immune checkpoint inhibitors-induced immune mediated hepatitis reaches 14.5%. Since these patients usually develop into liver failure, it is urgent to find out a more suitable therapy. Artificial liver support system (ALSS) treatment has been proved to effectively control both immune mediated hepatitis and liver failure, it may be a new therapy for immune checkpoint inhibitors-induced liver failure (ICIs-LF) in patients with HCC. Therefore, this study aims to investigate the efficacy and safety of ALSS treatment, including the classic mode of plasma exchange (PE) and new combination mode of double plasma molecular adsorption system (DPMAS) with sequential low-dose plasma exchange (LPE), for ICIs-LF in patients with HCC. Sixty patients with HCC and ICIs-LF will be enrolled in this study. The participants are randomly divided into trial group (DPMAS+LPE, and comprehensive internal medical treatment) and control group (PE and comprehensive internal medical treatment). Symptoms, signs, laboratory tests results, adverse events, mortality rates are recorded from treatment baseline to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 65 years old;
2. Clinical diagnosis of chronic hepatitis b virus infection (positive hepatitis b surface antigen or positive hepatitis b virus DNA > 0.5 year);
3. Clinical diagnosis of hepatocellular carcinoma and receive immune checkpoint inhibitors treatment. The last treatment of immune checkpoint inhibitors is less than three months from inclusion;
4. The level of hepatitis b virus DNA < 2000 IU/mL；
5. Serum aspartate aminotransferase/alanine aminotransferase > 20 times upper limit of normal；serum total bilirubin>10 times upper limit of normal；
6. Prothrombin time international ratio > 1.5;
7. Platelets > 50*10 E9/L;
8. Without intrahepatic bile duct dilation due to tumor progression.

Exclusion Criteria:

1. Other active liver diseases;
2. Other malignancy;
3. Pregnancy or lactation;
4. Human immunodeficiency virus infection or congenital immune deficiency diseases;
5. Severe diabetes, autoimmune diseases; unstable infarction due to cardio-cerebrovascular events; other important organ dysfunctions or transplantation;
6. Active bleeding, disseminated intravascular coagulation, thrombosis, or thrombotic disease;
7. Patients received artificial liver support system treatment in one week before inclusion;
8. Patients can not follow-up;
9. Investigator considering inappropriate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | 12 weeks
  Mortality rate at 12-week follow-up.

SECONDARY OUTCOMES:
Model for end-stage liver disease (MELD) score variation | 12 weeks
  Variation of MELD score at 12 weeks after treatment. MELD score = 9.57 × loge(creatinine mg/dl) + 3.78 × loge(TBIL mg/dl) + 11.20 × loge(PT-INR) + 6.43.

CONTACTS AND LOCATIONS:
Overall Officials: Wenxiong Xu, Doctor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, results and conclusions of this clinical trial will be published at academic conferences or in journals.
Supporting Information: Study Protocol, CSR
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Proposals should be directed to xuwenx@mail.sysu.edu.cn. To gain access, data requestors will need to sign a data access agreement

REFERENCES:
- [Derived] Luo Q, Zhang Y, Li Z, Chen J, Deng Z, Lai J, Chen X, Xie C, Peng L, Liu Y, Xu W. Efficacy and safety of artificial liver support system treatment for immune checkpoint inhibitors related liver failure in patients with hepatocellular carcinoma: Protocol for a randomized controlled clinical trial. Heliyon. 2024 Oct 9;10(20):e39095. doi: 10.1016/j.heliyon.2024.e39095. eCollection 2024 Oct 30. PMID 39640621